CLINICAL TRIAL: NCT06969742
Title: Development and Clinical Application of Intervention Program to Improve Mental Health and Quality of Life of Pediatric Solid Tumor Survivors and Caregivers, a Multicenter, Experimental Group, Pre-and-post Evaluation Intervention Study
Brief Title: Development and Application of Intervention Program to Improve Mental Health and Quality of Life of Solid Tumor Survivors and Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Seoul National University Hospital (Other); Tree and Forest Psychological Counseling Center (Unknown)
Responsible Party: Principal Investigator, Joo-Young Kim, Principal Investigator, Senior Researcher, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NCC2024-0006; RS-2023-CC139231 (Other Grant/Funding Number: Ministry of Health and Welfare, Republic of Korea)
Record Dates: First submitted 2025-03-10; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Pediatric Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Experimental Group_After cancer treatment (Experimental): Patients and primary caregivers(guardians) who have completed the cancer treatment and the treatment end date is within 2 years, and who are randomized into a experimental group.
  This group undergoes 10 sessions of psycho-education and psychological intervention(7 core sessions and 3 elective sessions) which last approximately 40 to 50 minutes per session.
  The experimental group will carry out psychological questionnaires three times: before beginning the session, after the core session(7th session), and after the end of the whole session(10th session).
  Psychological questionnaires includes emotional behavior evaluation tools for patients and caregivers and family evaluation tools for caregivers.
  The experimental group will carry out neurocognitive assessments before beginning the session.
  Interventions: Other: Psycho-education and Psychological intervention_After cancer treatment
- Control Group_After cancer treatment (Other): Patients and primary caregivers(guardians) who have completed the cancer treatment and the treatment end date is within 2 years, and who are randomized into a wait list control group.
  This group waits for 7 weeks before engaging in the counseling sessions. This group undergoes the same sessions as the experimental_after cancer treatment group(10 sessions).
  The wait list group will carry out psychological questionnaires three times: after the enrollment, 7 weeks after the enrollment, and 10 weeks after the enrollment.
  Psychological questionnaires includes emotional behavior evaluation tools for patients and caregivers and family evaluation tools for caregivers.
  The wait list group will carry out neurocognitive assessments after the enrollment.
  Interventions: Other: Psycho-education and Psychological intervention_After cancer treatment
- Experimental Group_In cancer treatment (Experimental): Patients and primary caregivers(guardians) going through cancer treatment and who are randomized into a experimental group.
  This group undergoes 5 sessions of psycho-education and psychological intervention(4 core sessions and 1 elective sessions) which last approximately 40 to 50 minutes per session.
  The experimental group will carry out psychological questionnaires two times: before beginning the session, and after the core session(4th session).
  Psychological questionnaires includes emotional behavior evaluation tools for patients and caregivers and family evaluation tools for caregivers.
  The experimental group will carry out neurocognitive assessments before beginning the session.
  Interventions: Other: Psycho-education and Psychological intervention_In cancer treatment
- Control Group_In cancer treatment (Other): Patients and primary caregivers(guardians) going through cancer treatment and who are randomized into a wait list control group.
  This group waits for 4 weeks before engaging in the counseling sessions. This group undergoes the same sessions as the experimental_in cancer treatment group(5 sessions on psycho-education and psychological intervention; 4 core sessions and 1 elective sessions).
  The wait list group will carry out psychological questionnaires two times: after the enrollment, and 4 weeks after the enrollment.
  Psychological questionnaires includes emotional behavior evaluation tools for patients and caregivers and family evaluation tools for caregivers.
  The wait list group will carry out neurocognitive assessments after the enrollment.
  Interventions: Other: Psycho-education and Psychological intervention_In cancer treatment

INTERVENTIONS:
Other: Psycho-education and Psychological intervention_After cancer treatment — The intervention program consists of Psycho-education and Psychological intervention that includes cognitive behavioral therapy sessions and interventions for patients and caregivers.
  It integrates and applies various evidence-based theories; mindfulness theory, solution-focused theory, resilience theory, and family intervention theory.
  The intervention is divided into two sessions; core sessions and elective sessions. The after cancer treatment group undergoes 7 core sessions and 3 elective sessions, a total of 10 sessions.
  The sessions are conducted 1:1, either face-to-face or remote, and 1 to 2 times a week, approximately 50 minutes per session.
  Arms: Control Group_After cancer treatment; Experimental Group_After cancer treatment
Other: Psycho-education and Psychological intervention_In cancer treatment — The intervention program consists of Psycho-education and Psychological intervention that includes cognitive behavioral therapy sessions and interventions for patients and caregivers.
  It integrates and applies various evidence-based theories; mindfulness theory, solution-focused theory, resilience theory, and family intervention theory.
  The intervention is divided into two sessions; core sessions and elective sessions.
  The intervention is divided into two sessions; core sessions and elective sessions. The in cancer treatment group undergoes 4 core sessions and 1 elective session, which is selected out of the given three topics, a total of 5 sessions.
  The sessions are conducted 1:1, either face-to-face or remote, and 1 to 2 times a week, approximately 50 minutes per session.
  Arms: Control Group_In cancer treatment; Experimental Group_In cancer treatment

SUMMARY:
The research team will assess the psychological abilities like cognitive(how you think and figure things out) and psycho-social(the well-being at the intersection of the internal workings and external experience) functions of young patients who are diagnosed with solid tumor and their primary caregivers. After assessing the psychological abilities, the research team will provide counseling and educational sessions developed by the team. The sessions are provided on a 1:1 basis to each of the participants to verify whether the sessions helped to improve the quality of life, including mental health.

DETAILED DESCRIPTION:
This study targets pediatric and adolescent cancer patients who are in the acute-transitional survival period(during cancer treatment to within 2 years of treatment end date) and their primary caregivers. Evaluation on the cognitive and psycho-social functions of pediatric and adolescent patients and their primary caregivers are conducted beforehand. Subsequently, the patients and caregivers are provided with psycho-education and psychological intervention program developed by the research team. The program is provided on a 1:1 basis to each subject to verify its effectiveness in improving quality of life, including mental health.

For patients and caregivers starting or undergoing cancer treatment, the purpose and information of the study will be informed when they visit the research participating institution: National Cancer Center or Seoul National University Hospital. For patients and caregivers who have completed the cancer treatment and the treatment end date is within 2 years, the research team will screen the patients during the relevant period. The purpose and information of the study will be provided during outpatient treatment. The research involves vulnerable subjects such as minors, therefore under the consent of the caregiver(a legal guardian), consent form with age-appropriate explanations of the study will be provided.

Before beginning the session, the patients will carry out neurocognitive assessments. The assessments includes Intelligence (Korean Wechsler Intelligence Scale for Children 4th and 5th Edition/Korean Wechsler Intelligence Scale 4th Edition), Memory(Rey-Kim Memory Test), Executive Function(Kims Frontal-Executive Neuropsychological Test), Attention(Children's Color Trails Test, Advanced Test of Attention / Trail Making Test, Continuous Performance Test), and Visual-Motor Integration 6th Edition.

During the pre-evaluation and orientation session, a counseling structure is establish for the next sessions of the program. The psycho-education and psychological intervention program is developed by comprehensively reflecting patient and caregiver interviews, previous research, and research team opinions. The program integrates and applies various evidence based theories, such as mindfulness theory, solution-focused theory, resilience theory, and family intervention theory. Consisting of core modules and elective modules, the program varies whether the patient is starting or undergoing cancer treatment, or have completed the cancer treatment. For patients and caregivers starting or undergoing cancer treatment, 4 core sessions and 1 elective session(selected out of the provided 3 topics) will be conducted. For patients and caregivers whose treatment end date is within 2 years, 7 core sessions and 3 elective sessions will be conducted. Every session is a 1:1 basis except for the family session, which the patient and the caregiver will participate together. Each session will last approximately 40-50 minutes, and conducted 1-2 times a week. The psycho-education and psychological intervention program is provided by the participating research institution and research team who have participated in the development of the program: National Cancer Center, Seoul National University Hospital, and Tree and Forest Psychological Counseling Center. Each of the institution has an assigned clinical psychologist who will conduct the sessions of the program. The program can be conducted in person or remotely. For patients starting or undergoing treatment, an independent counseling room will be provided by the research participating institution conducting the cancer treatment. For those who live far away or have difficulty in traveling to participate the program, an online video platform (ZOOM) can be utilized, or the sessions can be conducted on an individual location requested by the research subject under agreement.

To verify the effectiveness of the program, the patients and caregivers will carry out psychological questionnaires 2~3 times, depending on the group they are randomized in. For patients and caregivers starting or undergoing treatment and randomized into experimental group(Experimental Group_In cancer treatment) will carry out the questionnaires 2 times: before beginning the session, and after the core session(4th session). For patients and caregivers starting or undergoing treatment but randomized into control group(Control Group_In cancer treatment) will also carry out the questionnaires 2 times: after enrollment, and 4 weeks after the enrollment. For patients and caregivers whose treatment end date is within 2 years and randomized into experimental group(Experimental Group_After cancer treatment) will carry out the questionnaires 3 times: before beginning the session, after the core session(7th session), and after the end of the whole session(10th session). For patients and caregivers whose treatment end date is within 2 years but randomized into control group(Control Group_After cancer treatment) will also carry out the questionnaires 3 times: after enrollment, 7 weeks after the enrollment, and 10 weeks after the enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 10 and 24, and diagnosed with pediatric solid tumor, who are undergoing treatment or survivors who have completed the treatment and the treatment end date is within 2 years.
* Parent or legal guardian who is a primary caregiver to children and adolescent patient of acute-transitional phase.
* Those whose cognitive ability is capable of verbal counseling and who agrees to the evaluation assessment.

Exclusion Criteria:

* Those who disagree to participate as a research subject.
* Those whose psycho-emotional state requires professional treatment or medical conditions precludes intervention.
* Those undergoing treatment and children and adolescent survivors of acute-transitional phase, whose prior intelligence assessment FSIQ score is less than 70. However, if the GAI score is 70 or higher, participation is possible after the principal investigator's interview, with linguistic competence taken into consideration.

Elimination Criteria:

* Those who withdraw consent of this research.
* Those who have difficulty participating due to worsening of disease or decease of patient.

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference between quality of life, before and after the psycho-education and psychological intervention: A comparison on pediatric solid tumor survivors | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  The quality of life of pediatric solid tumor survivor is measured by the following scale.
  Pediatric Quality of Life Inventory Version 4.0 - Korean (PedsQL)
  * The scale is a self-report questionnaire, designed to assess quality of life in people with acute and chronic health conditions across four dimensions: physical, emotional, social, and functional well-being.
  * The scale is administered to pediatric solid tumor survivors, age between 10 to 24, who are under going treatment or who have completed the treatment and the treatment end date is within 2 years.
  * It's a 5-point scale, range of 0 to 92, with higher scores indicating lower quality of life in patients.
The difference between quality of life, before and after the psycho-education and psychological intervention: A comparison on caregivers | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  The quality of life of caregiver is measured by the following scale.
  Caregiver Quality of Life Index-Cancer Korea Version(CQOLC-K)
  * The scale is designed to measure the quality of life of caregivers of patients in hospice care.
  * The scale is a self report questionnaire, administered to the caregivers.
  * It's a 5-point scale, range of 0 to 140, with higher scores indicating lower quality of life.
The difference between depression, before and after the psycho-education and psychological intervention: A comparison on pediatric solid tumor survivors | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  The depression of pediatric solid tumor survivor is measured by the following scale.
  Korean Children's Depression Inventory 2nd Edition(K-CDI-2)
  * The scale is designed to measure pediatric depression across 4 dimensions: negative mood/physical symptoms, feeling of low self-esteem, inefficiency, and interpersonal relationships.
  * The scale is a self-report questionnaire, administered to patients aged between 10-18.
  * It's a 3-point scale, evaluated using T-score, with 60-64 indicating a need for attention on depression, 65-69 indicating more attention on depression, and 70 or more, a very elevated score, indicating a lot of attention on depression.
The difference between depression, before and after the psycho-education and psychological intervention: A comparison on pediatric solid tumor survivors | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  The depression of pediatric solid tumor survivor is measured by the following scale.
  Korean Beck Depression Inventory 2nd Edition(K-BDI-2)
  * The scale is a self-report questionnaire, designed to measure depression in adults.
  * Administered to patients aged between 19-24, it's a 4-point scale, range of 0-63, with 14-19 indicating mild depression, 20-28 indicating moderate depression, 29-63 indicating severe depression.
The difference between depression, before and after the psycho-education and psychological intervention: A comparison on caregivers | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  The depression of caregiver is measured by the following scale.
  Korean Beck Depression Inventory 2nd Edition(K-BDI-2)
  * The scale is a self-report questionnaire, designed to measure depression in adults.
  * Administered to caregivers, it's a 4-point scale, range of 0-63, with 14-19 indicating mild depression, 20-28 indicating moderate depression, 29-63 indicating severe depression.

SECONDARY OUTCOMES:
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years. | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life, the following scales will be used.
  The quality of life of pediatric solid tumor survivor is measured with Pediatric Quality of Life Inventory Version 4.0 - Korean (PedsQL).
  The quality of life of caregivers is measured with Caregiver Quality of Life Index-Cancer Korea Version(CQOLC-K).

OTHER OUTCOMES:
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 10-18) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 10 to 18, the Pediatric Functional Assessment of Cancer Therapy-Br(Peds FACT-Br) will be used.
  The scale is a self-report questionnaire, designed to measure physical, emotional, social and family well-being of pediatric brain cancer patients between the ages of 7-18.
  It's a 5-point Likert scale, with higher score indicating lower quality in life.
  The scale will be administered only to brain tumor patients and survivors.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 10-18) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 10 to 18, the Korean Revised Children's Manifest Anxiety Scale 2nd Edition(K-RCMAS-2) will be used.
  The scale is a self-report questionnaire, designed to measure anxiety in children and adolescents ages between 10-18, across four dimensions: physical anxiety, worry, social anxiety, and performance anxiety.
  It's a 2-point scale(Yes or No), with higher score indicating higher level of anxiety, which will be interpreted as lower quality in life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 10-18) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 10 to 18, the Korean Children's Depression Inventory 2nd Edition(K-CDI-2) will be used.
  The scale is a self-report questionnaire, designed to measure pediatric depression in children and adolescents, ages between 7-17, across 4 dimensions: negative mood/physical symptoms, feeling of low self-esteem, inefficiency, and interpersonal relationships.
  It's a 3-point scale, with higher score indicating higher level of pediatric depression, which will be interpreted as lower quality in life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 10-18) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 10 to 18, the Youth Self Report(YSR) will be used.
  The scale is a self-report questionnaire, designed to measure problem behaviors and clinical problems of children and adolescents, ages between 10-18.
  It's a 3-point scale, with higher score indicating higher level of problem behaviors, which will be interpreted as lower quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 10-18) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 10 to 18, the Fear of Progression Questionnaire for Children(FoP-Q-SF/C) will be used.
  The scale is a self-report questionnaire, designed to measure progression of chronic illness related fear in children and adolescents between the ages of 10-18.
  It's a 5-point scale, with higher score indicating higher level of fear on progression of cancer, which will be interpreted as lower quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 10-18) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 10 to 18, the Executive Function Difficulty Screening Questionnaire(EFDSQ) will be used.
  The scale is a self-report questionnaire, designed to measure executive dysfunction in children and adolescents, ages of 6-18, across 4 dimensions: planning-organizing difficulties, behavior control difficulties, emotion control difficulties, and inattention.
  It's a 3-point scale, with higher score indicating higher level of functional difficulties, which will be interpreted as lower quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 10-18) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 10 to 18, the Resilience Scale for Youth(RS-Y) will be used.
  The scale is a self-report questionnaire, designed to measure resilience in children and adolescents, ages of 10-18, across 7 dimensions: self-efficacy, optimism, perseverance, interpersonal relationship, emotional regulation, independence, and support.
  It's a 3-point scale, with higher score indicating higher level of resilience, which will be interpreted as higher quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 10-18) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 10 to 18, the Treatment Compliance(developed by the research team) will be used.
  It's a self-report single question scale, asking whether he or she follows the doctor's or hospital's instructions well, from 0(not compliant to instructions) to 10(comply to instructions) It's administered to children, adolescents, and young adults between the ages of 10-24, with higher score indicating higher compliance, which will be interpreted as higher quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 10-18) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 10 to 18, the Pediatric Functional Assessment of Cancer Therapy-Br(Peds FACT-Br) will be used.
  The scale is a caregiver-report questionnaire, designed to measure physical, emotional, social and family well-being of pediatric brain cancer patients, ages between 7-18.
  It's a 5-point Likert scale, with higher score indicating lower quality in life.
  The scale will be administered only to pediatric brain tumor patient's and survivor's caregivers.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 10-18) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 10 to 18, the Pediatric Quality of Life Inventory Version 4.0(PedsQL) will be used.
  The scale is a caregiver-report questionnaire, designed to assess quality of life in patients with acute and chronic health conditions across four dimensions; physical, emotional, social, and functional well-being.
  The scale is a 5-point scale, with higher score indicating lower quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 10-18) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 10 to 18, the Child Behavior Checklist 6-18(CBCL 6-18) will be used.
  The scale is a caregiver-report questionnaire, designed to measure problem behaviors and clinical problems of children and adolescents ages between 6-18.
  It's a 3-point scale, with higher score indicating higher level of problem behaviors, which will be interpreted as lower quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 10-18) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 10 to 18, the Korean ADHD Rating Scale(K-ARS) will be used.
  The scale is a caregiver-report questionnaire, designed to measure problems related to ADHD in children and adolescents, ages between 5-17.
  It's a 4-point Likert scale, with higher score indicating higher level of hyper activities, attention deficit, and impulsivity, which will be interpreted as lower quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 10-18) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 10 to 18, the Executive Function Difficulty Screening Questionnaire(EFDSQ) will be used.
  The scale is a caregiver-report questionnaire, designed to measure executive dysfunction in children and adolescents, ages 6-18, across 4 dimensions: planning-organizing difficulties, behavior control difficulties, emotion control difficulties, and inattention.
  It's a 3-point scale, with higher score indicating higher level of functional difficulties, which will be interpreted as lower quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 10-18) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 10 to 18, the Treatment Compliance(developed by the research team) will be used.
  It's a caregiver-report single question scale, asking whether the caregiver thinks the patient follows the doctor's or hospital's instructions well, from 0(not compliant to instructions) to 10(comply to instructions).
  Higher score indicates higher compliance, which will be interpreted as higher quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 19-24) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 19 to 24, the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Brain Neoplasm 20(EORTC QLQ-BN20) will be used.
  The scale is a self-report questionnaire, designed to measure health-related quality of life of patients with brain tumor.
  It's a 4-point Likert scale, with higher score indicating lower quality of life.
  The scale will be administered only to pediatric brain tumor patients and survivors.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 19-24) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 19 to 24, the Korean-Beck Depression Inventory 2nd Edition(K-BDI-2) will be used.
  The scale is a self-report questionnaire, designed to measure depression in adults.
  It's a 4-point scale, with higher score indicating higher level of depression, which will be interpreted as lower quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 19-24) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 19 to 24, the Korean-Beck Anxiety Inventory(K-BAI) will be used.
  The scale is a self-report questionnaire, designed to measure anxiety in adults.
  It's a 4-point Likert scale, with higher score indicating higher level of anxiety, which will be interpreted as lower quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 19-24) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 19 to 24, the Adult Self Report(ASR) will be used.
  The scale is a self-report questionnaire, designed to measure problem behaviors and clinical problems in adults between the ages of 19-59.
  It's a 3-point scale, with higher score indicating higher level of problem behaviors, which will be interpreted as lower quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 19-24) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 19 to 24, the Resilience Scale(RS) will be used.
  The scale is a self-report questionnaire, designed to measure resilience in adults across 7 dimensions: self-efficacy, optimism, perseverance, interpersonal relationship, emotional regulation, independence, and support.
  It's a 3-point scale, with higher score indicating higher level of resilience, which will be interpreted as higher quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 19-24) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 19 to 24, the Treatment Compliance(developed by the research team) will be used.
  It's a self-report single question scale, asking whether he or she follows the doctor's or hospital's instructions well, from 0(not compliant to instructions) to 10(comply to instructions).
  It's administered to children, adolescents, and young adults between the ages of 10-24, with higher score indicating higher compliance, which will be interpreted as higher quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 19-24) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 19 to 24, the Pediatric Quality of Life Inventory Version 4.0(PedsQL) will be used.
  The scale is a caregiver-report questionnaire, designed to assess quality of life in patients with acute and chronic health conditions across four dimensions: physical, emotional, social, and functional well-being.
  The scale is a 5-point scale, with higher score indicating lower quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 19-24) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 19 to 24, the Adult Behavior Checklist(ABCL) will be used.
  The scale is a caregiver-report questionnaire, designed to obtain information from people who know the adult(in this case, the patient): spouses, parents, siblings and friends.
  It's a 3-point scale, with higher score indicating higher level of problem behaviors, which will be interpreted as lower quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: A comparison between survivors starting/undergoing treatment, and survivors whose treatment end date is within 2 years (ages of 19-24) | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life for patients ages between 19 to 24, the Treatment Compliance(developed by the research team) will be used.
  It's a caregiver-report single question scale, asking whether the caregiver thinks the patient follows the doctor's or hospital's instructions well, from 0(not compliant to instructions) to 10(comply to instructions).
  Higher score indicates higher compliance, which will be interpreted as higher quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: intervention in caregivers | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life of caregivers, the Emotional Stress Inventory(ESI) will be used.
  The scale is a self-report questionnaire, designed to measure emotional stress, such as anger, anxiety, and depression, in both state and trait aspects in adults between the ages of 18-65.
  It's a 6-point Likert scale, with higher score indicating higher level of stress, which will be interpreted as lower quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: intervention in caregivers | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life of caregivers, the Korean-Beck Anxiety Inventory (K-BAI) will be used.
  The scale is a self-report questionnaire, designed to measure anxiety in adults.
  It's a 4-point Likert scale, with higher score indicating higher level of anxiety, which will be interpreted as lower quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: intervention in caregivers | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life of caregivers, the Fear of Progression Questionnaire for Parents of children with cancer(FoP-Q-SF/PR) will be used.
  The scale is a self-report questionnaire, designed to measure progression of chronic illness related fear in parents of pediatric cancer patients.
  It's a 5-point scale, with higher score indicating higher level of fear on progression of cancer, which will be interpreted as lower quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: intervention in caregivers | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life of caregivers, the Perceived Stress Scale(PSS) will be used.
  The scale is a self-report questionnaire, designed to measure the perception of stress in adults.
  It's a 5-point Likert scale, with higher score indicating higher level of perceived stress, which will be interpreted as lower quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: intervention in caregivers | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life of caregivers, the Parenting Sense of Competence(PSOC) will be used.
  The scale is a self-report questionnaire, designed to measure confidence and satisfaction in parenting and interest in their children.
  It's a 5-point Likert scale, that measure across 3 dimensions; efficacy, satisfaction, and interest.
  Higher score indicates lower level of satisfaction and interest in parenting, which will be interpreted as lower quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: intervention in caregivers | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life of caregivers, the Family Communication Scale Korean(FCS-K) will be used.
  The scale is a self-report questionnaire, designed to measure the communication level and pattern in family.
  It's a 5-point Likert scale, with higher score indicating higher level of effective family communication, which will be interpreted as higher quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: intervention in caregivers | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life of caregivers, the Family Adaptability and Cohesion Evaluation Scale 4th Edition(FACE-4) will be used.
  The scale is a self-report questionnaire, designed to measure family adaptability and family cohesion.
  It's a 5-point Likert scale, with higher score indicating higher level of adaptability and cohesion, which will be interpreted as higher quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: intervention in caregivers | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life of caregivers, the A Short Form of Post-Traumatic Growth Inventory(PTGI-SF) will be used.
  The scale is a self-report questionnaire, designed to measure positive changes after post-traumatic experience.
  It's a 6-point scale, with higher score indicating higher level of positive change, which will be interpreted as higher quality of life.
Correlation between intervention stages of psychological intervention program and improvement in quality of life: intervention in caregivers | After cancer treatment groups' intervention takes approximately 10 weeks, in cancer treatment groups' intervention takes approximately 5 weeks.
  To analyze the correlation between intervention stages and quality of life of caregivers, the Resilience Scale(RS) will be used.
  The scale is a self-report questionnaire, designed to measure resilience in adults across 7 dimensions; self-efficacy, optimism, perseverance, interpersonal relationship, emotional regulation, independence, and support.
  It's a 3-point scale, with higher score indicating higher level of resilience, which will be interpreted as higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — National Cancer Center; Co-Investigator, Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - National Cancer Center, Goyang-si, Gyonggi-do
  - Tree and Forest Psychological Counseling Center, Seoul, Seoul
  - Seoul National University Children's Hospital, Seoul, Seoul

IPD SHARING:
Plan to Share IPD: No